CLINICAL TRIAL: NCT00097604
Title: Valerian for Sleep Disturbance in Healthy Older Adults
Brief Title: Effects of Valerian on Sleep in Healthy Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Carol A. Landis, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26241-D; R21AT002108-01 (NIH); 04-2201-D 01 (Other: University of Washington Human Subjects Division)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2009-12

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep; Aged; Valerian; Complementary Therapies; Medicine, Herbal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valerian (Experimental): This study used a cross-over design with valerian compared to placebo. Group 1 received valerian first followed by placebo after washout and cross-over; group 2 received placebo first followed by placebo after wash-out and cross-over.
  Interventions: Dietary Supplement: Valerian root extract
- Placebo (Placebo Comparator): This study used a cross-over design with valerian compared to placebo. Group 1 received valerian first followed by placebo after washout and cross-over; group 2 received placebo first followed by placebo after wash-out and cross-over.
  Interventions: Dietary Supplement: Valerian root extract

INTERVENTIONS:
Dietary Supplement: Valerian root extract — Valerian root extract, 100 mg softgels, 3 softgels each night for 2 weeks, 30 minutes before bedtime
  Other Names: Valerian

SUMMARY:
The purpose of this study is to examine the way valerian, an herbal sleep agent, is absorbed and distributed in the body. This study will also compare the effects of valerian after 1 week versus after 2 weeks.

DETAILED DESCRIPTION:
Sleep disturbances are common among the elderly and may increase the risk for depression and early mortality. Use of over-the-counter sleep aids may disrupt sleep patterns and have serious side effects. Herbal medicines have the potential to improve sleep quality. Evidence suggests that valerian may improve sleep with a low rate of side effects, but its efficacy has not been thoroughly examined in the elderly. This study will determine the effectiveness and pharmacokinetics (PK) of valerian in older adults who experience disturbances in their sleep.

This study will last 8 weeks. At the sleep clinic, participants will be randomly assigned to receive either valerian or placebo on the first night of study enrollment. Participants will have an intravenous (IV) line inserted into their arms and multiple blood draws will be taken during their sleep for PK studies. The next day, participants will be sent home for a drug wash-out period and will return after 1 week for a 3-night stay at the clinic on Nights 8, 9, and 10. On Night 8, participants will adjust to their surroundings and begin a sleep log to describe the quality of their sleep; they will continue to note observations on their sleep in the sleep log for the duration of the study. Recordings of each participant's sleeping and breathing patterns will be taken on Nights 8 and 9 to screen for sleep disorders. On Night 10, participants will again be randomly assigned to receive either valerian or placebo. After Night 10, participants will be sent home and asked to continue taking their assigned intervention nightly for 11 nights. Participants will be asked to continue their sleep logs and begin a symptom log describing insomnia symptoms. After 11 nights, participants will return for another 3-night stay at the clinic on Nights 22, 23, and 24; participants will receive either valerian or placebo. Participants will then be sent home for a 12-day drug wash-out period; participants will return to the clinic for Nights 37 and 38. Night 37 will be an adaptation night; on Night 38, participants will be given the intervention they were not yet assigned on Night 24. After Night 38, participants will be asked to go home and continue their second treatment for 11 nights; participants will come back to the sleep clinic for another 3-night stay on Nights 50, 51, and 52 for observation and PK studies. After Night 52, participants will be sent home and asked to continue their sleep and symptoms logs for two more nights, then mail the logs to study researchers for analysis.

During this study, participants will be asked to keep logs of the quality of their sleep and of the insomnia symptoms they may be experiencing. In addition to the logs, post-sleep interviews will be used to assess the quality of participants' sleep and the number of awakenings. Participants' heart and breathing rates and leg movements will be measured during their stays at the sleep clinic. Participants will also have an activity monitoring device attached to either their wrist or waist for most of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pittsburgh Sleep Quality Instrument score higher than 5
* Insomnia Severity Index score less than 22
* At least 5 years past menopause, for female participants

Exclusion Criteria:

* Current use of prescribed or over-the-counter sleep medications
* Plans to move from the area within 2 months of study entry
* Significant signs and symptoms of sleep apnea; periodic leg movements in sleep (PLMS) associated with arousals; rapid eye movement (REM) behavior disorder; restless legs syndrome; advanced sleep phase syndrome; delayed sleep phase syndrome; or any other sleep disorder, including severe insomnia or a history of chronic insomnia, for which standard therapy would be the treatment of choice
* Shift work within 6 months prior to study entry
* Current unusual or highly unstable sleep schedule
* Trans-meridian travel across more than three time zones within 4 weeks prior to study entry
* Body mass index between 18 kg/m2 and 32 kg/m2
* Significant and uncontrolled major illness or psychiatric disease
* Cognitive impairment
* Current life stress
* Use of tobacco within 6 months prior to study entry
* Excessive use of alcohol or caffeine
* Currently taking hormone replacement therapy hypnotic or psychotropic medication

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Landis, DNSc, Principal Investigator — University of Washington, School of Nursing
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Taibi DM, Vitiello MV, Barsness S, Elmer GW, Anderson GD, Landis CA. A randomized clinical trial of valerian fails to improve self-reported, polysomnographic, and actigraphic sleep in older women with insomnia. Sleep Med. 2009 Mar;10(3):319-28. doi: 10.1016/j.sleep.2008.02.001. Epub 2008 May 14. PMID 18482867